CLINICAL TRIAL: NCT06616025
Title: Phase 3, Multicenter, Randomized, Subject and Evaluator Blinded, Controlled Study Evaluating the Safety and Efficacy of NTX-001 Compared to Standard of Care (Neurorrhaphy) in the Treatment of Upper Extremity Transected Nerves Requiring Surgical Repair.
Brief Title: This Study Will Evaluate the Effectiveness of NTX-001, a Surgical Nerve Repair Product When Used in People With Upper Extremity Nerve Lacerations.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Neuraptive Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NTx24301
Record Dates: First submitted 2024-09-24; First posted 2024-09-27 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-03

CONDITIONS: Peripheral Nerve Injury Upper Limb; Peripheral Nerve Injury (PNI)
Keywords: Transected Nerves; Requiring Surgical Repair; Upper Extremity
MeSH Terms: conditions — Peripheral Nerve Injuries

STUDY DESIGN:
Intervention Model Description: Treatment vs. Standard of Care
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: All study personnel involved in the surgical procedure will be unblinded. Patient, Care Providers and outcomes evaluators will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- NTX-001 (Experimental): NTX-001 used during the surgical repair of an upper extremity peripheral nerve injury in conjunction with standard suture neurorrhaphy.
  Interventions: Combination Product: NTX-001 (PEG-Fusion)
- Standard Suture Neurorrhaphy (No Intervention): Standard of Care

INTERVENTIONS:
Combination Product: NTX-001 (PEG-Fusion) — One time use surgical product, 3 solutions applied topically, in sequence, to the peripheral nerve repair site, in conjunction with standard suture neurorrhaphy.
  Arms: NTX-001

SUMMARY:
NTX-001 is a single use surgical product intended for use in conjunction with standard suture neurorrhaphy of severed nerves in patients between 18 and 80.

DETAILED DESCRIPTION:
NTX-001 has been developed as a surgical product to be used in conjunction with standard suture neurorrhaphy of a severed nerve. Use of NTX-001 is intended to safely accelerate the often slow and diminished return of function in repaired nerves. It often takes months and/or years to determine if function will be restored. By that point, restoration is often incomplete and can result in lifelong motor and/or sensory deficits. By reconnecting (PEG-fusion) a substantial number of axons within a severed nerve, the degeneration-regeneration cycle and subsequent atrophy may be reduced or even prevented for those axons and their targets, respectively. NTX-001 (PEG-fusion) has the potential to avoid the consequences of protracted denervation of distal target tissues by eliminating the period of total denervation thus reducing the time to stable recovery and providing greater innervation to affected tissues.

ELIGIBILITY:
Inclusion Criteria:

* The subject has voluntarily agreed to participate in this study and has signed an Institutional Review Board (IRB) approved informed consent form.
* The subject is between eighteen (18) and eighty (80) years of age.
* The subject has clinical evidence of a Sunderland's 4th degree (Class II) or 5th degree (Class III) nerve transection(s) that has resulted in upper extremity nerve impairment that requires surgical treatment.

Exclusion Criteria:

* Subjects whose nerve repair will occur greater than 48 hours after nerve transection.
* Subjects requiring nerve repair involving an autograft, allograft or conduit(s).
* Subjects with multiple transected nerve injuries are allowed into the study only if all injuries are amenable to direct repair.
* Subjects who, in the judgement of the investigator, are not likely to demonstrate meaningful recovery within a reasonable time frame during follow up due to significant muscle atrophy or other morbidity.
* The subject's injury is a result of a suicide attempt or self- harm.
* The subject has documented history or clinical signs of any condition where NTX-001 might not prove beneficial (e.g., systemic neuromuscular disease, systemic neurological deficit, or other treatments known to affect the growth and/or physiology of the neural and vascular system).
* The subject has a known allergy to polyethylene glycol (PEG) or human grade silicone.
* The subject is pregnant or breastfeeding.
* The subject is currently enrolled in another investigational study or has participated in an investigational study within 30 days prior to screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Mean Michigan Hand Questionnaire (MHQ) Two Domain Score (ADL and Pain) | Screening Visit, Week 24
  The Activities of Daily Living component evaluates the ability to perform specific tasks using either hand or both hands together. The Pain subdomain addresses the frequency and intensity of pain in both the right and left hands/wrists, along with its impact on sleep and daily activities, and the emotional distress it causes. The raw scale score for each of the 6 scales is the sum of the responses of each scale item. The raw score is converted to a score range from 0 to 100. 100 being the best.

SECONDARY OUTCOMES:
Intraoperative CheckPoint® Stimulation. | In Operating Room
  A CheckPoint® Stimulator will be used intra-operatively to detect immediate reconnection of severed peripheral nerves (axons) in mixed-motor nerves only. The measures include in response of direct nerve stimulation, proximally and distally to suture site.
Electromyography (EMG) Testing | Weeks 12, 24.
  EMG will be used to detect reconnection of severed peripheral nerves (axons) using PEG Fusion. Restoration of nerve conduction indicates the restoration of axon continuity, which is a prerequisite for the prevention for Wallerian degeneration, neuromuscular junction degeneration, muscle atrophy and functional recovery.
Nerve Conduction Velocity (NCV) | Weeks 12, 24
  NVC testing measures how fast an electrical impulse moves through a nerve.
MHQ Total Score | Weeks 2, 4, 6, 8, 10, 12, 16, 20, 24, 30, 36, 42, and 48
  The MHQ quantifies different impairments between the subjects in uninjured and involved upper extremities. A general survey of hand function includes twenty-five items for the right and the left hand, as well as questions for both hands. Questions regarding function specifically refer to the impact of the involved hand and/or wrist on the activity which presumably takes all joints of the upper extremity into account. The overall questionnaire is scored from 0 to 100, with 100 being the optimal score.
Time to Return to Function | Screening Visit, Weeks 2, 4, 6, 8, 10, 12, 16, 20, 24, 30, 36, 42, and 48.
  Achievement of seventy-five (75)% function in the combined ADL and pain MHQ domain scores. The Activities of Daily Living component evaluates the ability to perform specific tasks using either hand or both hands together. The Pain subdomain addresses the frequency and intensity of pain in both the right and left hands/wrists, along with its impact on sleep and daily activities, and the emotional distress it causes. The overall questionnaire is scored from 0 to 100, with 100 being the optimal score.
Change in NPRS | Screening Visit, Weeks 2, 4, 6, 8, 10, 12,16, 20, 24, 30, 36, 42, and 48
  The NPRS is used to assess for pain and to determine pain intensity. The NPRS is an 11-point scale scored from 0-10: 1) "0" = no pain 2) "10" = the most intense pain imaginable. The average of the 3 ratings is used to represent the subject's level of pain over the previous 24 hours.
Semmes Weinstein Monofilament Test (SWMT) | Weeks 2, 4, 8, 12, 24, 36, 48.
  SWMT provides information on protective sensation, the rigorous system can detect relatively minor differences in sensory function, and changes will occur early in nerve injury. The assessment tool consists of a set of monofilaments that vary in thickness and diameter, the gradient forces of these monofilaments that subjects' can feel, range from 0.086 gm to 0.448gm. The normal value in the hand is in the range of the green filament (1.65 to 2.83 mN).
MHQ Two Domain Score | Weeks 2, 4, 6, 8, 10, 12, 16, 20, 30, 36, 42, 48
  The Activities of Daily Living component evaluates the ability to perform specific tasks using either hand or both hands together. The Pain subdomain addresses the frequency and intensity of pain in both the right and left hands/wrists, along with its impact on sleep and daily activities, and the emotional distress it causes. The raw scale score for each of the 6 scales is the sum of the responses of each scale item. The raw score is converted to a score range from 0 to 100. 100 being the best.
Change from Week 2 in MHQ Two Domain Score | Weeks 2, 4, 6, 8, 10, 12, 16, 20, 24, 30, 36, 42, and 48.
  The Activities of Daily Living component evaluates the ability to perform specific tasks using either hand or both hands together. The Pain subdomain addresses the frequency and intensity of pain in both the right and left hands/wrists, along with its impact on sleep and daily activities, and the emotional distress it causes. The raw scale score for each of the 6 scales is the sum of the responses of each scale item. The raw score is converted to a score range from 0 to 100. 100 being the best.
Medical Research Council Classification (MRCC) Sensory Score | Weeks 2, 4, 8, 12, 24, 36, and 48.
  The scale is commonly used including 2 Point Discrimination for grading the sensory outcome after peripheral nerve surgery. This scale is categorized into S0-S4: S0 is the absence of sensibility; S1 is the recovery of deep cutaneous pain; S2 is the return of superficial cutaneous pain and some degree of tactile sensibility; S3 is the return of superficial cutaneous pain and tactile sensibility without over response; and S4 is the complete recovery.
Medical Research Council Classification (MRCC) Motor Score | Weeks 2, 4, 8, 12, 24, 36, 48
  This assessment is conducted on mixed motor nerve injuries only. Strength can best be assessed by isolating an individual muscle group and comparing power with that of the subject. It can be conducted to assess larger muscles or muscle groups as well as intrinsic muscles of the hand. Measuring the difference between the affected limb and the contralateral limb. 0/5 is no muscle activation whatsoever; 1/5 is muscle activation without limb movement; 2/5 implies that the limb can be moved only when gravity is taken out of the equation; 3/5 means that the subject can overcome gravity but not resistance;• 4/5 (or 4+ or 4-) implies weakness with enough strength to overcome varying degrees of physical resistance; 5/5 is full strength.
Columbia-Suicide Severity Rating Scale | Screening Visit, Weeks 4, 12 and 48
  The Columbia-Suicide Severity Rating Scale (C-SSRS) is a unique suicide risk assessment tool that supports suicide risk assessment. The answers identify whether someone is at risk for suicide, assessing the severity and immediacy of that risk, and gauging the level of support that the person needs. Based on the answers to the questions, the score determines if the subject is at a low, medium, or high risk for suicide.
Change from Baseline (W2) in Numeric Pain Rating Scale (NPRS) | Weeks 2, 24.
  The NPRS is used to assess for pain and to determine pain intensity. The NPRS is an 11-point scale scored from 0-10: 1) "0" = no pain 2) "10" = the most intense pain imaginable. The average of the 3 ratings is used to represent the subject's level of pain over the previous 24 hours.
Patient Global Impression of Change Score | Weeks 2, 4, 6, 8, 10, 12, 16, 20, 30, 36, 42, and 48
  This scale evaluates all aspects of patients; health and assesses if there has been an improvement or decline in clinical status. PGIC is a 7-point scale depicting a subjects rating of overall improvement. The subject rates their change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse."
Change in Total MHQ Score | Weeks 2, 4, 6, 8, 10, 12, 16, 20, 24, 30, 36, 42, and 48.
  The MHQ quantifies different impairments between the subjects uninjured and involved upper extremities. It was designed as a general survey of hand function and includes twenty-five items for the right and the left hand, as well as questions for both hands. Furthermore, questions regarding function specifically refer to the impact of the involved hand and/or wrist on the activity which presumably takes all joints of the upper extremity into account. The overall questionnaire is scored from 0 to 100, with 100 being the optimal score.
Patient Global Impression of Change Score (PGIC) | Week 24
  This scale evaluates all aspects of subjects health and assesses if there has been an improvement or decline in clinical status. PGIC is a 7-point scale depicting a subjects rating of overall improvement. The subject rates their change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse."

CONTACTS AND LOCATIONS:
Overall Officials: Seth Schulman, MD, Study Director — Neuraptive Therapeutics Inc.
Locations (7):
- United States (7):
  - Orlando Health Orlando Regional Medical Center, Orlando, Florida
  - University of Chicago, Chicago, Illinois
  - Curtis National Center at MedStar Union Memorial Hospital, Baltimore, Maryland
  - Missouri Orthopaedic Institute, Columbia, Missouri
  - Barnes-Jewish Hospital 1 Barnes Jewish Hospital Plaza St., St Louis, Missouri
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Harborview Medical Center, Seattle, Washington

REFERENCES:
- See also: Sponsor Website — https://www.neuraptive.com/